CLINICAL TRIAL: NCT01760798
Title: To Compare Efficacy of Weekly Versus Daily Teriparatide in the Management of Postmenopausal Osteoporosis
Brief Title: Weekly vs Daily Teriparatide Therapy in Severe Postmenopausal Osteoporosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Sanjay K. Bhadada, Associate Professor, Dept of Endocrinology, Post Graduate Institute of Medical Education and Research, Chandigarh
Organization: PIMERIndia (Unknown)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: teriparatide
Record Dates: First submitted 2013-01-02; First posted 2013-01-04 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-04

CONDITIONS: Osteoporosis
Keywords: osteoporosis; Teriparatide
MeSH Terms: conditions — Osteoporosis | interventions — Teriparatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Daily Teriparatide group (Active Comparator): This group will recieve 20µg of teriparatide by subcutaneous route daily at 8 pm for 1 year
  Interventions: Drug: Teriparatide
- Weekly Teriparatide group (Experimental): This group will recieve 60µg of teriparatide by subcutaneous route weekly at 8pm on Sunday for 1 year
  Interventions: Drug: Teriparatide

INTERVENTIONS:
Drug: Teriparatide

SUMMARY:
Osteoporosis is characterized by decreased bone strength and it is prevalent among postmenopausal women but also occurs in men and women with underlying conditions or major risk factors associated with bone demineralization. Its chief clinical manifestations are vertebral and hip fractures, although fractures can occur at any skeletal site.The World Health Organization (WHO) operationally defines osteoporosis as a bone density that falls 2.5 standard deviations (SD) below the mean for young healthy adults of the same gender-also referred to as T-score of -2.5. Postmenopausal women who fall at the lower end of the young normal range (a T-score of >1 SD below the mean) are defined as having low bone density (osteopenia) and are also at increased risk of osteoporosis. More than 50% of the fractures, including hip fractures, among postmenopausal women occur in this group.

Teriparatide is one of the most effective treatment options for osteoporosis. But the cost of teriparatide is prohibitively expensive and in countries like India with limited personal resources of the individuals, its not a feasible option in the majority of the patients with severe osteoporosis. The investigators aim to compare weekly versus daily teriparatide therapy in an open label non inferiority trial and if successful, the investigators anticipate, the cost of treatment could be reduced considerably so that treatment becomes more affordable to a larger number of patients. Also with weekly therapy, number of multiple injections could be brought down.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women of age group 50-70 having T score less than -2.5 SD or lower at lumbar spine or proximal femur.

Exclusion Criteria:

* Patients with renal dysfunction (serum creatinine >1.5)
* Primary and secondary hyperparathyroidism
* Secondary osteoporosis
* Unexplained elevated ALP (alkaline phosphatase)
* History of therapeutic radiation
* Active malignancy and patients having implant
* Patients who have received i.v. or oral bisphosphonates in their disease course

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-06 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
BMD at Hip and lumber spine | 1 year
  DEXA scan(BMD at hip and lumbar spine) at baseline and at the end of 1 year
Reduction in fracture risk | 6 week, 6 month and 1 year
  Reduction in fracture risk using online FRAX tool( WHO fracture risk assessment tool) at baseline and at 1year

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Kr Bhadada, DM, Principal Investigator — Associate Professor, Department of Endocrinology, PGIMER Chandigarh India
Locations (1):
- PGIMER, Chandigarh, Uttarakhand, India